CLINICAL TRIAL: NCT05877313
Title: Phase 2a Multicenter, Randomized, Double-Blinded, Placebo-Controlled Clinical Trial To Evaluate The Safety And Efficacy Of Topical Nitric Oxide Releasing Solution For The Treatment Of Human Papillomavirus Verrucae Plantaris
Brief Title: Nitric Oxide Releasing Solution (NORS) For The Treatment Of Human Papillomavirus(HPV) Verrucae Plantaris (Plantar Warts)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanotize Research and Development corp. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HPV-Warts-01
Record Dates: First submitted 2023-05-06; First posted 2023-05-26 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Verruca Plantaris
Keywords: Plantar Warts; Warts; HPV
MeSH Terms: conditions — Warts | interventions — Nitric Oxide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Nitric Oxide Releasing Solution 1X (Active Comparator): Foot bath with nitric oxide releasing solution (NORS) at 1X dosage delivered 3 times weekly (Mon, Wed, Fri).
  500mL NORS in a footbath @ 4110 ppm*min
  Interventions: Drug: Nitric Oxide
- Nitric Oxide Releasing Solution 2X (Active Comparator): Foot bath with nitric oxide releasing solution (NORS) at 2X dosage delivered 3 times weekly (Mon, Wed, Fri).
  500mL NORS in a footbath @ 12190 ppm*min
  Interventions: Drug: Nitric Oxide
- Vehicle Control (Placebo Comparator): Foot bath with sterile water delivered 3 times weekly (Mon, Wed, Fri)
  500mL sterile water in a foot bath.
  Interventions: Other: Sterile water foot bath

INTERVENTIONS:
Other: Sterile water foot bath — Participants will use the same foot bath and sterile water used in the treatment arm minus the active ingredients.
  Arms: Vehicle Control
Drug: Nitric Oxide — Participants will use a foot bath filled with 500mL of NORS for 15 min. The solution's two components are mixed 1:1 to 500mL in the foot bath immediately before treatment. The solution contains NO at 68.9ppm*hrs and 203.2ppm*hrs for 1X and 2X solutions respectively, and it acts as a virucidal agent. Instructions for storage, handling, and use will be provided to site staff and participants.
  Other Names: Nitric Oxide Releasing Solution (NORS)
  Arms: Nitric Oxide Releasing Solution 1X; Nitric Oxide Releasing Solution 2X

SUMMARY:
A phase 2a multicenter, randomized, double-blinded, placebo-controlled clinical trial to evaluate the safety and efficacy of topical nitric oxide releasing solution (NORS) for the treatment of human papillomavirus (HPV) caused verrucae plantaris (plantar warts). Participants will be treated over a 21 day period with a final evaluation on Day 35. They will be separated into 3 treatment groups (placebo, 1x and 2x dose). Participants will be evaluated for change in wart size, wart clearance, and HPV genotype.

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blinded, placebo-controlled phase 2a clinical trial to evaluate the safety and efficacy of NORS in adolescent and adult volunteers as a treatment for verrucae plantaris (plantar warts). Participants aged 12 or older with plantar warts on the bottom of the foot (feet) will be enrolled into one of 3 cohorts in a ratio of 1:1:1 (NORS1X, 3 doses/week; NORS 2X, 3 doses/week; placebo vehicle, 3 doses/week for 3 weeks).

Participants with or without underlying medical conditions (unless exclusionary) seeking treatment at the site for plantar warts will be eligible. Eligible recruited participants will have three or more currently active plantar warts on the bottom of their foot/feet. Participants who are currently pursuing other forms of treatment (e.g., over-the-counter wart removers, a treatment recommended by their physician, or are waiting for a current treatment) will be excluded from the study.

After enrollment and randomization participants will self-administer study treatment--defined as either blinded study NORS footbath treatment, or placebo vehicle (sterile water) footbath treatment--three times a week for three weeks. Study treatment will be delivered via a single footbath filled with 500 mL of NORS solution. Placebo treatment will be delivered via a single footbath filled with 500 mL of vehicle solution. Each treatment will be a 15-minute soaking time per foot. If both feet are affected, the participant will receive the same treatment on both feet. Thirty (30) participants will be enrolled, with 10 participants per treatment. The study duration is five weeks, which includes Screening/Baseline (Day 0), 3 weeks (21 days) of Treatment, and 14 days of Follow-Up. Lesions will be scored at enrollment (Day 0) and subsequently at follow-up visits (Day 7, Day 14, Day 21, Day 28, and Day 35).

The primary endpoint is to evaluate the efficacy of NORS to provide lesion clearance by photographic lesion length measurement (Day 35). Photographs and counting of warts will be performed at each visit. Wart length and clearance evaluation will be recorded at each site visit to Day 35. Lesion clearance is defined as a length of 0 mm. After each wart assessment (at site visits), warts may be debrided, as necessary per the investigators' evaluation and standard of care. Secondary endpoints will assess lesions for the mean reduction in dimensions as measured by the change in longest length size from baseline observed at Days 7, 14, 21, 28, and 35; lesion clearance by Physician Wart Assessment (PWA=0); and pain reduction using an 11- point Pain Numeric Rating Scale (NRS; 0 to 10), An exploratory endpoint will evaluate the distribution of HPV genotypes determined by swabbing the overlaying skin of the wart from participants at baseline. Participants will additionally have their vitals tracked and skin visually assessed for inflammation at baseline (Day 0) and follow-up visits (Day 35). Adverse events will also be tracked as a measure of safety. The discontinuation rate for tolerance (unless for a lack of perceived efficacy) will also be tracked.

Participants will have six on-site visits. Screening and randomization will be completed on Day 0 followed by a three-week (21-day) treatment period (until Day 21). A site visit will occur on Day 7, Day 14, and at the end-of-treatment (EOT) site visit on Day 21. The treatment period will be followed by a 14-day follow-up period, with a visit on Day 28 and an end-of-study (EOS) visit on Day 35. During the entire study, the participant will be instructed to keep a daily journal of observations to report to the site investigator at their visits, i.e., when they observed each lesion's clearance, new occurrences of lesions, or recurrence of the same lesions.

During the visits on Days 7, 14, 21, 28, and 35 (Follow-Up), the investigator/study staff will review and assess information about lesion clearance, pain, other outcomes, and/or adverse events. At the screening/baseline/randomization visit and at the EOT visit, the patient's medical history (including prior/concomitant illness, medication, adverse event), physical examination, and vital signs assessment will be conducted/recorded. Urine pregnancy tests will be conducted in women of childbearing potential at the screening visit and at EOT visit/early termination visit.

Data collection and monitoring will be performed remotely and on-site. Screening and enrollment will take place on-site with consenting procedure performed in-person on-site. Participants will receive study treatment directly from the site. No laboratory bloodwork assessments will be performed.

ELIGIBILITY:
Inclusion Criteria:

* At least 12 years old at the time of consent.
* Three or more plantar warts (single foot, or both feet).
* If female, be surgically sterile or post-menopausal (no menses for at least 12 months), or if of childbearing potential, must be using an acceptable method of contraception such as a combination estrogen/progestin hormonal contraceptive (oral or injected) for at least 1 month prior to Day 1, or such items as an intrauterine device (IUD), intrauterine system (IUS), transdermal hormonal implant, vaginal hormonal ring, or 2 forms of the following: diaphragm, cervical cap, patch, condom, spermicide, or sponge. Total abstinence is permitted. Local requirements will apply if local regulations deviate from the previously listed contraception methods to prevent pregnancy. In addition, females of childbearing potential must agree to continue to use their method of birth control for the duration of the study.
* If male, be surgically sterile, or agree to use appropriate contraception (latex condom with spermicide) when engaging in sexual activity and agree not to donate sperm for the duration of the study.
* Be in good health (i.e., no acute illnesses or hospitalizations within 30 days of the study start, no planned procedures during study participation, and no newly diagnosed chronic illnesses that are not deemed stable by the participant's primary care physician), in the opinion of the Investigator, based on medical history (i.e., absence of any clinically relevant abnormality) during Screening.
* Be able to understand and provide written informed consent.
* Must be willing and able to manage the self-treatment and attend on-site study visits.

Exclusion Criteria:

* Participants with acute illnesses or hospitalizations within 30 days of the study start, and/or planned procedures during study participation, and/or newly diagnosed chronic illnesses that are not deemed stable by the participant's primary care physician), based on Investigator assessment of medical history during Screening.
* Participants who are currently in another trial for the treatment of warts.
* Participants with any unhealed or newly obtained infection, wound, injury, or lesion on the foot the month prior to Screening.
* Participants who are immunosuppressed, immunodeficient, or are receiving any form of immunosuppression drug.
* Participants with any prior history of neuropathy.
* Participants who are receiving concomitant treatment of plantar warts (involving any form of therapy).
* Females who are breastfeeding, pregnant, or attempting to become pregnant.
* Participants who have conditions that participation is not in their best interest, i.e., hypersensitivity to the product's ingredients.
* Participants with a recent ulcer, tumor, or surgery performed on their foot within the previous month.
* Participants whose participation in the study, in the opinion of the Investigator, have a condition that would interfere with their ability to adhere to the protocol (e.g., participants who are mentally or neurologically disabled and who are considered not fit to participate in the study), interfere with the assessment of the investigational product, or compromise the safety of the participant or the quality of the data.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-08-02 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-04-12 (Actual)

PRIMARY OUTCOMES:
To evaluate the efficacy of NORS as a treatment for verrucae plantaris as measured by lesion clearance (Day 35). | 35 Days
  The efficacy of NORS as measured by the clearance of the wart(s) defined by a photographic lesion measurement of zero (0) length and as compared to a placebo treatment

SECONDARY OUTCOMES:
To assess the mean reduction in lesion dimensions as measured by the change in size from baseline observed at Day 7, 14, 21, 28 and 35. | 35 days
  Reduction in lesion (plantar wart) size measured in millimeters with each NORS dose as compared to reduction with placebo treatment. Measurement of the longest dimension will be recorded and the mean reduction in dimensions as measured by the change in size from baseline observed at Day 7, 14, 21, 28 and 35.
To assess by mean changes in size of lesion as measured by area at Days 7, 14, 21, 28 and 35 and lesion clearance (Day 35). | 35 days
  Changes in the size (area) of lesion from baseline will be measured on each visit.
To evaluate (median) time to pain reduction of lesion(s). | 35 days
  Number of participants who experience reduced pain in their lesions and the time to reduction. This will be scored on an 11-point Pain Numeric Rating Scale (NRS; 0 to 10). Lesions will be scored at enrollment, daily by participants, and subsequently on follow up visits (Day 7, 14, 21, 28 and 35).
To assess the safety and tolerability of NORS. | 35 days
  Number of participants who find the NORS treatment tolerable.

OTHER OUTCOMES:
Evaluate the distribution of HPV genotypes. | Baseline visit only
  HPV genotypes will be determined by swabbing the overlaying skin of the warts from participants at baseline. Analysis will be performed using a multiplex PCR reaction.
Evaluate lesion clearance using an alternative assessment instrument. | 35 days
  Lesion clearance will be evaluated by the Physician Wart Assessment tool (PWA=0 on Day 35).
Evaluate a dermatologic quality of life instrument. | 35 days
  Dermatology Life Quality Index (DLQI) (questions score change from baseline at Day 35)

CONTACTS AND LOCATIONS:
Overall Officials: Keith Moore, PHARMMD, Study Director — SaNOtize R&D Corp
Locations (3):
- Canada (3):
  - Achilles Foot Health Centre, Surrey, British Columbia
  - Spectrum Health, Vancouver, British Columbia
  - Pacific Derm, Vancouver, British Columbia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schumacher SA, Dugom L, Martins J, Leemhuis J, Teskey SJL, Moore K, Miller CC. Efficacy and safety of a topical nitric oxide-releasing solution (NORS) as a noninvasive treatment for plantar warts (verrucae plantaris). J Dermatolog Treat. 2026 Dec;37(1):2610918. doi: 10.1080/09546634.2025.2610918. Epub 2026 Jan 6. PMID 41493215